CLINICAL TRIAL: NCT06586450
Title: Effect of Low Level Laser Versus Interferential Current on Postmenopausal Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola Saad Ibrahim El-Naggar, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005317
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Low-Level Light Therapy; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low level laser group (Experimental): The participants will receive low level laser therapy and core stability exercises
  Interventions: Device: Low level laser therapy; Other: Core stability exercise
- Interferential current group (Experimental): The participants will receive interferential current and core stability exercises
  Interventions: Device: Interferential current; Other: Core stability exercise
- Core stability exercise group (Active Comparator): The participants will perform core stability exercises only
  Interventions: Other: Core stability exercise

INTERVENTIONS:
Device: Low level laser therapy — The participants will receive Low Level Laser on lumbo-pelvic region for 20 min/sessions,3 sessions / week for 12 weeks, with the following parameters: Wavelength: 808 nm, continuous mode, Output power: 160 mw, Penetration depth: 4 cm, Power density:0.16 J/cm2.
  Arms: Low level laser group
Device: Interferential current — All participants will receive interferential current on lumbopelvic region ( quadripolar technique) for 25 min/session, 3 sessions/week for 12 weeks, with the following parameters: carrier frequency of 4 KHZ and sweep frequency 95 HZ, intensity based on patient's tolerance without muscle contraction.
  Arms: Interferential current group
Other: Core stability exercise — The participants will perform core stability exercises for 15 min 3 time/week in the form of Prone Gluteal Squeezes, Pelvic Bridging, Curl Up Exercise, and Double Knee to Chest Stretching Exercises.

SUMMARY:
This study will be conducted to compare the effect of low-level laser and interferential current on postmenopausal low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is a major health problem affecting majority of the people at some point of their life.The prevalence of postmenopausal LBP is 32.4%. It has major implication for quality of life, such as limitation of daily activities and physiological stress, being one of the main causes of work absenteeism.

The prolonged use of NSAIDs is associated with cardiovascular, hepatic, and renal problems. Therefore, there is a need for emphasis on alternative methods of conservative treatment as non-pharmacological and non-invasive therapy to relieve postmenopausal LBP.

Low level laser has been proven to have an impact on postmenopausal LBP, through several mechanisms as (a) increased endogenous opioid neurotransmitter production ;(b)raised threshold to thermal pain and enhanced local blood circulation ; (c)increased oxygen consumption by accelerating the redox reaction rate of the electron respiratory chain of mitochondria ; (d) increased adenosine triphosphate (ATP) production at the cellular level ;(e) increased production of the anti-inflammatory cytokines.

Also, another non- invasive technique is the interferential current which is one of the existing electrotherapy treatments used to reduce pain and has been studied for its effectiveness in relieving LBP through its deeper penetration into the tissues.

So, this study will be conducted to provide new evidence and information about the efficacy of low-level laser versus interferential current on LBP in postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

• Sixty postmenopausal women (at least one year after stoppage menses).

* Their age will be ranged from 50 to 60 years.
* Their body mass index (BMI) will be less than 30 kg/m2.
* All of them suffer from chronic low back pain (at least 3 months).
* The score of pain will be 2 or more according to visual analogue scale (VAS).

Exclusion Criteria:

* Spinal fracture or any other neurological disorder.
* Lumbar disc herniation, degenerative joint diseases, or spondylolisthesis.
* BMI>30 kg/m2
* Gynecological Diseases as Chronic pelvic pain or genital prolapse.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 12 weeks
  The intensity of postmenopausal low back pain will be assessed using a visual analogue scale (VAS) for all participants in the three groups before and after treatment, which is a method of representing subjects' pain on a 10 cm linear scale. A score of 0 means " no pain" and 10 means " very high degree of pain
Lumbar flexion range of motion | 12 weeks
  The modified Schober test will be used to measure the lumbar flexion range of motion (ROM) by using the tape measurement. Each participant will be asked to stand erect with her feet about shoulder-width apart to stabilize the pelvis. Then, the posterior superior iliac spines(PSIS) will be determined by the therapist's both thumbs, and then an ink line will be drawn along the midline of the lumbar spines horizontal to the PSIS to mark the midpoint between the two PSIS. Then tape will be used to identify and mark two points: one is 10 cm superior to the midpoint (A), and another is 5 cm inferior to the midpoint (B). The participant will be instructed to bend forward as much as she can while keeping both knees straight, the new distance between superior and inferior skin marking will be measured in centimeters. The increased distance along the tape due to lumbar flexion is normally about 6-7 cm (less than 5 cm should be considered abnormal).
Lumbar extension range of motion | 12 weeks
  The modified Schober test will be used to measure the lumbar extension range of motion (ROM) by using the tape measurement while the patient is in a standing position. The participant will be instructed to put her hands on her buttocks and bend backward into full lumbar extension and the new distance between the superior and inferior skin markings will be measured in centimeters by the tape measurement. The change in the difference between the marks is used to indicate the amount of lumbar extension. The increased distance along the tape due to the extension of the lumbar spine is normally about 2-3 cm (less than 1cm should be considered abnormal).
Lumbar lateral flexion range of motion | 12 weeks
  The participant will be asked to stand erect with her feet about shoulder-width apart. Both right and left lateral flexion will be measured by the tape as the distance from the tip of the index finger to the floor at maximal comfortable lateral flexion. The participant will be instructed to bend her trunk laterally as much as she can. The normal value of lateral spinal flexion is 16.2-28.0 cm.

SECONDARY OUTCOMES:
Functional disability | 12 weeks
  Functional disability will be assessed by the Oswestry Disability Index, it was developed as a clinical valid and reliable assessment tool that would provide an estimate of disability expressed as a percentage score. It is composed of 10 questions and it takes around 5min for a patient to complete. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, bed-bound. A low score = low degree of disability, a high score = high degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Azza B Kassab, professor, Study Chair — Cairo University
Locations (1):
- Ola Saad El Naggar, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol